CLINICAL TRIAL: NCT07165964
Title: Nursing Interventions to Enhance Positive Mental Health and Self Care in Women During the Climacteric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Marta Prats Arimon, Co-Investigador, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003099 JORDI GOL; CER032510 (Other Grant/Funding Number: Ministerio de Igualdad. Spanish Goverment)
Record Dates: First submitted 2025-08-12; First posted 2025-09-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09

CONDITIONS: Climacteric Symptoms; Climactericum; Self Care
Keywords: climateric symptoms; women; climactericum; self care; positive mental health

STUDY DESIGN:
Intervention Model Description: Model pre-post test in intervention group and pre-post usual follow up in control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Climateric Intevention Group (IG) (Active Comparator): Intervention Group (IG):
  Participants will complete the same pre- and post-intervention assessments, including the validated scales and the ad hoc instrument used in the study.
  Participants in the intervention group will receive a personal access code to a Moodle virtual campus, where they will find a series of specially designed podcasts and videos addressing self-care during the climacteric and promoting positive mental health (PMH). These digital resources-referred to as "digital pills"-have been developed by experts in the field to meet the specific needs of this population.
  Each resource will be followed by a brief quiz to assess participant engagement, knowledge acquisition, and adherence. At the end of the intervention, participants will also complete a satisfaction survey. Access to the platform will remain open for two months, during which participants can view the materials and complete the quizzes at their own pace, alongside receiving usual care.
  Interventions: Behavioral: Personal interventions in Climateric
- Control Group (CG) (No Intervention): Control Group (CG):
  Participants in the control group will complete the same pre- and post-intervention assessments, including the validated scales and the ad hoc instrument used in the study. The intervention for this group will consist of routine follow-up care provided by a midwife in primary care, focusing on the management of climacteric symptoms. No additional digital resources or structured educational content will be provided beyond standard care.

INTERVENTIONS:
Behavioral: Personal interventions in Climateric — The intervention group (IG) will participate in the climacteric care program. Each participant will receive a personal access code to a Moodle-based virtual campus, where they will find specially designed podcasts and videos, provided in addition to standard care. These digital "pills" have been developed by subject matter experts to support self-care during the climacteric stage and to promote positive mental health (PMH). Each resource is followed by a short quiz to assess engagement, knowledge acquisition, and adherence. A final satisfaction survey will also be included. IG participants will have two months of access to explore the content, complete the quizzes, and interact with the platform.
  The intervention includes the following modules:
  MODULE 1: INTRODUCTION TO THE CLIMACTERIC/MENOPAUSE MODULE 2: DIETARY HABITS AND PHYSICAL ACTIVITY MODULE 3: PSYCHOEMOTIONAL MANAGEMENT
  Arms: Climateric Intevention Group (IG)

SUMMARY:
This study will test whether a nursing program using podcasts and videos can help women feel better and take better care of themselves during the climacteric (the stage leading up to and following menopause). Women between 42 and 58 years old who attend public sexual and reproductive health clinics in the Metropolitan South Health Region of Barcelona (Sant Boi, Sant Feliu, and Cornellà) will be invited to participate.

Participants will be randomly assigned to one of two groups:

Intervention Group: will receive access to podcasts and videos offering practical advice and strategies to improve emotional well-being and self-care.

Control Group: will receive standard care. All participants will complete questionnaires before and after the program to assess symptoms, mental health, and satisfaction with self-care. Statistical methods will be used to compare the results between both groups and determine whether the program produces a significant difference.

The aim of the study is to demonstrate that this digital nursing intervention is effective and could be implemented more broadly in healthcare settings.

DETAILED DESCRIPTION:
Self-Care and Positive Mental Health During the Climacteric Stage: Conceptual Framework and Social Relevance

Self-care is a fundamental human function, particularly vital during the climacteric stage, when women experience significant physical, emotional, and social changes. The conceptual foundation of this project is Dorothea Orem's General Theory of Self-Care Deficit, which encompasses both the individual's capacity for self-care and their ability to care for others. Orem defines self-care as "the personal actions undertaken and performed by each individual to maintain life, health, and well-being, and to consistently respond to their health needs."

Despite the importance of this life stage, the scientific literature indicates that most interventions targeting health issues in women during the climacteric have been non-holistic, often addressing physical and emotional aspects in isolation. There is a notable lack of empirical evidence supporting interventions that simultaneously promote self-care and positive mental health (PMH) in menopausal women. Existing studies tend to focus on problem-solving strategies, lifestyle modifications, and empowerment programs aimed at improving quality of life. However, no specific programs have been identified that address PMH in this population.

Both PMH and self-care capacity are essential constructs for women adapting to the multifaceted changes of the climacteric. Enhancing these dimensions may contribute significantly to health promotion during this extended phase of the female life cycle, which is often marked by conditions that negatively impact quality of life. Research suggests that psychosocial factors such as optimism, emotional stability, and self-esteem are positively associated with well-being and resilience. Moreover, several studies support a bidirectional relationship between self-care and PMH, indicating that improvements in one domain can reinforce the other. A notable example is the PiPsE program, which aims to enhance PMH in individuals with chronic illnesses.

The outcomes of this project are expected to advance the field of women's health by deepening our understanding of the needs of women during the menopausal transition, particularly in relation to PMH and self-care. These findings may inform the development of tailored intervention programs that support women's health across all stages of menopause, aligning with broader health promotion and disease prevention policies.

This proposal aligns with Strategic Line DEM.2.2.4 of the III Strategic Plan for Effective Equality of Women and Men (2022-2025), which advocates for "the implementation of sexual and reproductive health programs at all life stages." By addressing the menopausal stage-a period often overlooked in empirical research-this project contributes to a more comprehensive understanding of women's health. Furthermore, incorporating a gender perspective in health research is essential to correcting and eliminating gender biases in the diagnosis, treatment, and conceptualization of women's physiological and psychological processes. This study promotes a positive, health-affirming approach to women's physical and mental well-being, centering the voices of menopausal women as primary stakeholders.

Utility and Relevance for Social Sectors

This innovative project reorients the focus of women's sexual health from the reproductive phase to its conclusion-menopause-during which women undergo a range of physical, psychoemotional, and social transformations. It is imperative that society recognize and value the resilience and strength of women in this stage, beyond their reproductive roles. Accordingly, this project seeks to highlight women's psychoemotional capacities, self-care abilities, and the broader social significance of these attributes.

It is also essential to provide women with platforms to articulate their physical and emotional needs throughout the climacteric (pre-, peri-, and post-menopause). The findings of this study should inform the design of programs that promote PMH, emotional well-being, and self-care capacity within a health promotion framework, empowering women to take an active role in managing their health. Additionally, this research will help define a distinct domain of women's health, separate from the male sexual and reproductive trajectory.

Evidence continues to show that caregiving responsibilities disproportionately fall on women. As highlighted in the Research Team Experience section, who has long been committed to strengthening the physical and mental resilience of women caregivers through initiatives that promote PMH and self-care. During menopause, many women also assume caregiving roles for elderly dependents, which can exacerbate the physical and emotional challenges of this life stage. This underscores the urgent need to support and reinforce women's self-care-both physical and mental-during the climacteric.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 42-58 years attending the participating ASSIR centers.
* Clinically identified symptoms of climacteric during routine consultation.

Exclusion Criteria:

* Cognitive or learning impairments preventing comprehension of study procedures.
* Physical, emotional, or intellectual limitations hindering completion of study instruments or participation in the intervention.
* Current treatment for hormone dependent cancer.
* Use of an intrauterine device or ongoing hormonal contraceptives.
* Other medical causes of secondary menopause.

Ages: 42 Years to 58 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of positive mental health on 39 points of the Positive Mental Health Scale | Baseline and one month post-intervention
  The SMP multifactorial scale consists of 39 items that are distributed among 6 factors: Personal Satisfaction, Prosocial Attitude, Self-Control, Autonomy, Problem Solving and Self-Update, and Interpersonal Relationship Skills. The evaluation of each item is done with a scale scale ranging from 1 to 4. Being 1, always or almost always, 2, quite often, 3 often and 4, never or almost never. Finally, a score between 39 and 156 is obtained, the higher the score the more positive mental health.
Changes observed in the severity and number of symptoms within the somatic-vegetative, psychological, and urogenital domains during the climacteric. | Baseline and one month post-intervention
  The level of symptoms associated with the climacteric will be measured using the Menopause Rating Scale (MRS), a validated instrument that assesses the somatic-vegetative, psychological, and urogenital domains. The scale will be administered before and after the intervention to evaluate changes in symptom intensity across these domains.
Levels of self-care capacity will be assessed using a validated instrument: the Agency for Self-Care Assessment Scale | Baseline and one month post-intervention
  The Self-Care Agency Scale (ASA) (Evers and Isenberg, 1989) is a tool designed to assess an individual's overall capacity for self-care. The scale consists of 24 items (16 positive items and 8 negative items), with questions 2, 6, 11, 13, 14, 15, 20 and 23 reverse-scored for the purpose of analysis. The scale utilised is of a Likert-type design, incorporating four possible responses that are tallied for the purpose of analysis. The participants were asked to indicate their level of agreement or disagreement with the following statements using a scale of 1 to 4: 1 = Strongly Disagree, 2 = Disagree, 3 = Agree, 4 = Total Agreement. The results of this study range from 24 (minimum self-care ability) to 96 (maximum self-care ability), thus establishing a cut-off point of <48 to define low self-care ability.

CONTACTS AND LOCATIONS:
Overall Officials: Monsterrat Puig-Llobet, Principal Investigator — Universitat de Barelona
Locations (1):
- Universitat de Barceñpma, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD when the periode of collecting data is finished.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start in september 2025 until desember 2025
Access Criteria: All team researchers from University of Barcelona can share IPD throught SPSS program by corporative mail.All researchers need a password to access the institution's intranet. In addition, a shared folder will be generated where only researchers have access to share other documents.

REFERENCES:
- [Result] Puig Llobet M, Sanchez Ortega M, Lluch-Canut M, Moreno-Arroyo M, Hidalgo Blanco MA, Roldan-Merino J. Positive Mental Health and Self-Care in Patients with Chronic Physical Health Problems: Implications for Evidence-based Practice. Worldviews Evid Based Nurs. 2020 Aug;17(4):293-300. doi: 10.1111/wvn.12453. Epub 2020 Aug 6. PMID 32762130
- [Result] Wherry DC, Rob CG, Marohn MR, Rich NM. An external audit of laparoscopic cholecystectomy performed in medical treatment facilities of the department of Defense. Ann Surg. 1994 Nov;220(5):626-34. doi: 10.1097/00000658-199411000-00005. PMID 7979610
- [Result] Chen C. Assessment of myocardial viability in patients with chronic coronary disease. Circulation. 1997 Oct 21;96(8):2740-2. No abstract available. PMID 9355926
- [Result] Yamamoto T, Katayama I, Nishioka K. Involvement of basic fibroblast growth factor in fibroblast-stimulatory serum activity of a patient with systemic lupus erythematosus and multiple dermatofibromas. Dermatology. 1995;191(4):281-5. doi: 10.1159/000246569. PMID 8573922
- [Result] Khalil J, Boutros S, Kheir N, Kassem M, Salameh P, Sacre H, Akel M, Obeid S, Hallit S. Eating disorders and their relationship with menopausal phases among a sample of middle-aged Lebanese women. BMC Womens Health. 2022 May 10;22(1):153. doi: 10.1186/s12905-022-01738-6. PMID 35538474
- [Result] Kafaei-Atrian M, Sadat Z, Nasiri S, Izadi-Avanji FS. The Effect of Self-care Education Based on Self-efficacy Theory, Individual Empowerment Model, and Their Integration on Quality of Life among Menopausal Women. Int J Community Based Nurs Midwifery. 2022 Jan;10(1):54-63. doi: 10.30476/IJCBNM.2021.86814.1370. PMID 35005041
- [Result] Carr, A., Cullen, K., Keeney, C., Canning, C., Mooney, O., Chinseallaigh, E., & O'Dowd, A. (2021). Effectiveness of positive psychology interventions: A systematic review and meta-analysis. The Journal of Positive Psychology, 16(6), 749-769. https://doi.org/10.1080/17439760.2020.1818807